CLINICAL TRIAL: NCT02661321
Title: Location and Timing of Inhaler Use, Exacerbations and Physical Activity in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vincent S. Fan, Staff Physician, VA Puget Sound Health Care System
Other Study IDs: VA HSR&D PPO 10-299
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention was used in this study, this was an observational study

SUMMARY:
This was an observational pilot study to examine the usefulness of an electronic sensor that monitors short-acting beta-agonist inhaled medication use. The goals of this study were to: 1) test the feasibility of using the inhaler sensor to measure worsening symptoms and exacerbations, 2) characterize physical activity in patients with COPD, and 3) examine whether environmental factors can be linked to mild exacerbations measured by the inhaler sensor.

DETAILED DESCRIPTION:
Objectives: This study tested the usefulness of a GPS-enabled inhaler to study the associations between air pollution, chronic obstructive pulmonary disease (COPD) exacerbations, and physical activity. Specific aims are 1) test the feasibility of using the inhaler sensor to measure worsening symptoms and exacerbations, 2) characterize physical activity in patients with COPD, and 3) examine whether environmental factors can be linked to mild exacerbations measured by the inhaler sensor.

Research Design: A 12-week observational, longitudinal pilot study of patients with COPD.

Methodology: Participants recruited at VA Puget Sound performed spirometry and completed baseline questionnaires. An inhaler sensor was placed on their albuterol inhaler to record the time and location of inhaler actuation throughout the three month follow-up. Each month participants answered questions regarding their breathing symptoms and physical activity. Physical activity was measured by self-report using a weeklong Physical Activity Checklist. A pedometer was worn at three 7 day periods. Public use air pollution and meteorological data will be linked to the inhaler data. We will compute descriptive statistics for all measures, including sociodemographics, exacerbation rates, inhaler use, air pollution exposures and physical activity levels. In addition, a time series analysis will be used to test if the frequency of inhaler use is associated with higher levels of daily air pollution.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC<0.70
* FEV1 >30% and <FEV1<65% predicted
* Participants must be able to walk without assistance
* No plans to leave the study area during the 12-week study period
* Non-smoker and not live with someone who smokes
* No history of asthma
* Use a short-acting bronchodilator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease at VA Puget Sound Health Care System in Seattle, WA
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Exacerbations | 3 months
  Number of exacerbations during the 3-month follow-up period

SECONDARY OUTCOMES:
Physical activity: Total number of steps per day | Up to 3 months
  An Omron pedometer was used by patients for 7 days at baseline, week 4, week 10 during the 3 month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fan, MD MPH, Principal Investigator — VA Puget Sound HCS, Seattle, WA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sumino K, Locke ER, Magzamen S, Gylys-Colwell I, Humblet O, Nguyen HQ, Thomas RM, Fan VS. Use of a Remote Inhaler Monitoring Device to Measure Change in Inhaler Use with Chronic Obstructive Pulmonary Disease Exacerbations. J Aerosol Med Pulm Drug Deliv. 2018 Jun;31(3):191-198. doi: 10.1089/jamp.2017.1383. Epub 2017 Oct 16. PMID 29035120